CLINICAL TRIAL: NCT06013059
Title: A Comparative Study Between the Different Levels of TMJ Arthroscopy in the Management of TMJ Internal Derangement (A Randomized Clinical Trial)
Brief Title: A Comparative Study Between the Different Levels of TMJ Arthroscopy in the Management of TMJ Internal Derangement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Hamza Fayad, Assistant lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001056 - IORG 0008839
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: TMJ Disc Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- level (I) arthroscopy (Lysis and lavage) (Active Comparator)
  Interventions: Procedure: three levels of TMJ arthroscopy
- level (II) arthroscopy (operative arthroscopy) (Active Comparator)
  Interventions: Procedure: three levels of TMJ arthroscopy
- level (III) arthroscopy (operative arthroscopy + disc repositioning and fixation) (Active Comparator)
  Interventions: Procedure: three levels of TMJ arthroscopy

INTERVENTIONS:
Procedure: three levels of TMJ arthroscopy — Group I: 10 patients will be treated with Lysis and lavage
  Arms: level (I) arthroscopy (Lysis and lavage)
Procedure: three levels of TMJ arthroscopy — Group II: 10 patients will be treated with operative arthroscopy
  Arms: level (II) arthroscopy (operative arthroscopy)
Procedure: three levels of TMJ arthroscopy — Group III: 10 patients will be treated with operative arthroscopy + discopexy
  Arms: level (III) arthroscopy (operative arthroscopy + disc repositioning and fixation)

SUMMARY:
The temporomandibular joint (TMJ) arthroscopy has emerging role nowadays in the treatment of TMJ internal derangement with its three levels of intervention. A comparative study between the 3 levels is essential to develop a standardized selection criteria and management algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TMJ internal derangement Wilkes III

Exclusion Criteria:

1. Medically unfit patients.
2. Patients with TMDs secondary to malocclusion.
3. Psychological instability.
4. Patients operated before for other TMJ problems.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Mouth opening measurement | 1, 3 and 6 months postoperatively
  measuring the maximal interincisal opening (MIO)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Fayad, MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT06013059/Prot_SAP_ICF_000.pdf